CLINICAL TRIAL: NCT01050595
Title: Methylnaltrexone for the Reversal of Opiate-Induced Constipation in the Intensive Care Unit
Brief Title: Methylnaltrexone for Treatment of Opiate-Induced Constipation in the Intensive Care Unit
Acronym: MOVE-IT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. John Health System, Michigan (Other)
Responsible Party: Bradford Whitmer, DO, Providence Medical Center and Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 107199
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Opioid-induced Constipation
Keywords: Intensive Care Unit; Constipation; Bowel Management
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylnaltrexone Bromide (Active Comparator)
  Interventions: Drug: Methylnaltrexone Bromide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo-Normal Saline

INTERVENTIONS:
Drug: Methylnaltrexone Bromide — The experimental group will receive the recommended dose of MNTX (Relistor) is 8 mg for patients weighing 38 kg to less than 62 kg (84 lbs to less than 136 lbs) or 12 mg for patients weighing 62 kg to 114 kg (136 lbs to 251 lbs). Patients whose weight is below 38 kg or greater than 114 kg, will be dosed at 0.15 mg/kg. If creatinine clearance <30 will decrease dose by 50%. This will be given after 72 hours of no bowel movement. Bowel management protocol will be instituted four hours afterward with the methylnaltrexone being given every other day.
  Other Names: Relistor
  Arms: Methylnaltrexone Bromide
Drug: Placebo-Normal Saline — Control group will be given an equal amount of normal saline in an identically appearing vial every other day until a bowel movement occurs. A bowel management protocol will also be started.
  Other Names: Relistor
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if there will be a significantly higher incidence of a bowel movement with methylnaltrexone vs. placebo within 4 hours +- 45 minutes with decreased need for rescue medications in the intensive care unit in patients with opioid-induced constipation. Patients will also be managed with an aggressive bowel management protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older in the ICU
* Opioids for analgesia for at least 24 hours.
* Opioid-induced constipation with no bowel movement within the last 72 hours.
* Women of childbearing potential had negative pregnancy tests.

Exclusion Criteria:

* Contraindication to use of the GI tract
* Diarrhea on admission
* Bowel surgery within 8 weeks of admission
* Ileostomy or colostomy
* Not expected to live or stay more than 3 days in the intensive care unit
* Constipation that was not primarily caused by opioids (as determined by the investigator)
* No opioid use in the last 24 hours,
* Mechanical gastrointestinal obstruction
* An indwelling peritoneal catheter
* Clinically active diverticular disease
* Fecal impaction
* Acute surgical abdomen
* History of Crohn's disease or ulcerative colitis
* On Palliative care
* Less than 18 years old
* Bowel movement in last 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
A significantly higher incidence of a rescue free laxation with methylnaltrexone within 4 hours +- 45 minutes. | Nine months

SECONDARY OUTCOMES:
Decreased need for rescue medications to have a bowel movement in the treatment arm vs placebo. | Nine months

CONTACTS AND LOCATIONS:
Overall Officials: Bradford A Whitmer, D.O., Principal Investigator — Providence Hospital and Medical Center
Locations (1):
- Providence Hospital and Medical Center, Southfield, Michigan, United States

REFERENCES:
- [Background] Ritchie G, Burgess L, Mostafa S, Wenstone R. Preventing constipation in critically ill patients. Nurs Times. 2008 Nov 18-24;104(46):42-4. PMID 19054971
- [Background] Patanwala AE, Abarca J, Huckleberry Y, Erstad BL. Pharmacologic management of constipation in the critically ill patient. Pharmacotherapy. 2006 Jul;26(7):896-902. doi: 10.1592/phco.26.7.896. PMID 16803421
- [Background] Chappell D, Rehm M, Conzen P. Opioid-induced constipation in intensive care patients: relief in sight? Crit Care. 2008;12(4):161. doi: 10.1186/cc6930. Epub 2008 Jul 1. PMID 18598388
- [Background] Mostafa SM, Bhandari S, Ritchie G, Gratton N, Wenstone R. Constipation and its implications in the critically ill patient. Br J Anaesth. 2003 Dec;91(6):815-9. doi: 10.1093/bja/aeg275. PMID 14633751
- [Background] Tittle M, McMillan SC. Pain and pain-related side effects in an ICU and on a surgical unit: nurses' management. Am J Crit Care. 1994 Jan;3(1):25-30. PMID 7906992
- [Background] Viscusi ER, Gan TJ, Leslie JB, Foss JF, Talon MD, Du W, Owens G. Peripherally acting mu-opioid receptor antagonists and postoperative ileus: mechanisms of action and clinical applicability. Anesth Analg. 2009 Jun;108(6):1811-22. doi: 10.1213/ane.0b013e31819e0d3a. PMID 19448206
- [Background] Arpino PA, Thompson BT. Safety of enteral naloxone for the reversal of opiate-induced constipation in the intensive care unit. J Clin Pharm Ther. 2009 Apr;34(2):171-5. doi: 10.1111/j.1365-2710.2008.00982.x. PMID 19250137
- [Background] McKenna S, Wallis M, Brannelly A, Cawood J. The nursing management of diarrhoea and constipation before and after the implementation of a bowel management protocol. Aust Crit Care. 2001 Feb;14(1):10-6. doi: 10.1016/s1036-7314(01)80017-5. PMID 11899755
- [Background] Dorman BP, Hill C, McGrath M, Mansour A, Dobson D, Pearse T, Singleton J, Al-Omoush A, Barry M, Colongon AR, Perez M, Fitzgerald D, Zabala M. Bowel management in the intensive care unit. Intensive Crit Care Nurs. 2004 Dec;20(6):320-9. doi: 10.1016/j.iccn.2004.09.004. PMID 15567673
- [Background] Hill S, Anderson J, Baker K, Bonson B, Gager M, Lake E. Management of constipation in the critically ill patient. Nurs Crit Care. 1998 May-Jun;3(3):134-7. PMID 9883173
- [Background] Sanz Rubiales A, del Valle Rivero ML. Methylnaltrexone for opioid-induced constipation in advanced illness. N Engl J Med. 2008 Sep 4;359(10):1070-1; author reply 1071. doi: 10.1056/NEJMc081373. No abstract available. PMID 18768955